CLINICAL TRIAL: NCT01257802
Title: GnRH-a for Ovarian Protection During CYC Therapy for Rheumatic Diseases
Acronym: LUPRON
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Joseph Mccune (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Joseph Mccune, Michael H. and Marcia S. Klein Professor of Rheumatic Diseases and Director, Lupus Clinic, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00043071; 5R01HD066139 (NIH)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Lupus Erythematosus, Systemic; Systemic Vasculitis; Isolated Angiitis of Central Nervous System; Lung Disease With Systemic Sclerosis; Lung Disease Interstitial Diffuse
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Systemic Vasculitis | interventions — Leuprolide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LUPRON (Active Comparator): Monthly depot leuprolide acetate 3.75 mg injection during cyclophosphamide administration. First dose of study drug given at least 10 days before following dose of cyclophosphamide if cyclophosphamide is given in biweekly or monthly boluses
  Interventions: Drug: depot leuprolide acetate 3.75 mg
- Placebo (Placebo Comparator): Monthly placebo injection during cyclophosphamide administration. First dose of study drug given at least 10 days before following dose of cyclophosphamide if cyclophosphamide is given in biweekly or monthly boluses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: depot leuprolide acetate 3.75 mg — Monthly depot leuprolide acetate 3.75 mg vs placebo during cyclophosphamide administration. First dose of study drug given at least 10 days before following dose of cyclophosphamide if cyclophosphamide is given in biweekly or monthly boluses
  Other Names: LUPRON depot 3.75 mg
  Arms: LUPRON
Drug: Placebo — Monthly placebo during cyclophosphamide administration. First dose of study drug given at least 10 days before following dose of cyclophosphamide if cyclophosphamide is given in biweekly or monthly boluses
  Arms: Placebo

SUMMARY:
The purpose of this study it to determine whether the use of a gonadotropin releasing hormone (GnRH)-agonist (depot-leuprolide acetate) during cyclophosphamide (CYC) therapy in women with rheumatic diseases will provide greater ovarian protection than placebo.

DETAILED DESCRIPTION:
Patients will be women ages 18-40 with either a severe rheumatic disease requiring cyclophosphamide or interstitial lung disease requiring cyclophosphamide to be administered either daily orally; monthly intravenously; or intravenously every 2 weeks for 6 doses. Because cyclophosphamide treatment may be required urgently for some indications, study entry may occur before either the first or second dose of cyclophosphamide for patients receiving cyclophosphamide intravenously.

Of 16 participants who were screened, only 14 were randomized and only 7 participants actually completed the study. Due to this low number, follicle stimulating hormone (FSH) levels were not obtained.

Secondary outcome measures that are not available include presence of menses and FSH.

ELIGIBILITY:
1. Female, post menarche, not menopausal
2. Ages 18-40 years inclusive at enrollment
3. Diagnosis consistent with a rheumatic or autoimmune disease requiring 3-6 months of daily or intermittent cyclophosphamide therapy. This may include, but is not limited to:

   * Systemic lupus
   * Sjogren's syndrome
   * Systemic vasculitis
   * Isolated vasculitis of the central nervous system
   * Other autoimmune neurologic diseases requiring cyclophosphamide including transverse myelitis, peripheral neuropathies, multiple sclerosis, neuromyelitis optica, and retinal vasculitis
   * Behcet's syndrome
   * Scleroderma
   * Inflammatory myositis
   * Interstitial lung disease, other autoimmune pulmonary diseases requiring cyclophosphamide
   * Overlap connective tissue diseases not precisely fitting the above definitions clearly requiring cyclophosphamide for severe immune mediated organ damage
   * Rheumatoid vasculitis
4. Patients will have planned cyclophosphamide treatment according to any one of the following regimens:

   * 3 to 6 months of daily oral cyclophosphamide: Lupron/placebo must be given within four (4) weeks of initiation of daily cyclophosphamide.
   * The Eurolupus regimen consisting of 6 fortnightly biweekly boluses of 500 mg cyclophosphamide: First dose of Lupron/placebo must be given 10 days prior to the second dose of cyclophosphamide
   * 3 to 6 monthly boluses of cyclophosphamide by the NIH regimen: First dose of Lupron/placebo must be given 10 days prior to the second dose of cyclophosphamide
5. A satisfactory plan for contraception consistent with cyclophosphamide administration (when appropriate: depot progestins, IUD, combination oral contraception and/or dual barrier contraception).

Exclusion Criteria:

1. Symptoms consistent with ovarian failure based on gynecologic evaluation and confirmatory laboratory testing
2. Prior unilateral or bilateral oophorectomy
3. Cervical intraepithelial neoplasia (CIN 2, or more severe), that has not been adequately evaluated or is not being adequately treated
4. Contraindications to use of GnRH-a (e.g., undiagnosed abnormal uterine bleeding)
5. Prior adverse or allergic reaction to GnRH-a
6. A history of severe psychiatric disorders, particularly severe depression that is currently not adequately treated
7. History of significant noncompliance with medical treatment
8. Patients with major risk factors for decreased bone mineral content such as chronic alcohol and/or tobacco use, strong family history of osteoporosis, or chronic use of drugs that can reduce bone mass such as anticonvulsants that have not already been addressed with appropriate measures to preserve bone mass.
9. Pregnant or breastfeeding
10. Significant thrombotic event requiring treatment that will not have received appropriate therapy for at least 4 weeks before initiation of study drug.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J McCune, M.D., Principal Investigator — Professor of Internal Medicine
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 of the 16 consented individuals were screen fails and therefore were not randomized.
Groups:
- Placebo: depot leuprolide acetate 3.75 mg: Monthly depot leuprolide acetate 3.75 mg vs placebo during cyclophosphamide administration. First dose of study drug given at least 10 days before following dose of cyclophosphamide if cyclophosphamide is given in biweekly or monthly boluses
  Placebo: Monthly placebo during cyclophosphamide administration. First dose of study drug given at least 10 days before following dose of cyclophosphamide if cyclophosphamide is given in biweekly or monthly boluses
Period: Overall Study
Arm/Group | LUPRON | Placebo
Started | 6 | 8
6 Month / 24 Week Visit | 5 | 2
Completed | 5 | 2
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Population: Because only 14 people randomized, baseline data is provided for those for whom relevant outcome measures were achieved.
Groups:
- Total: Total of all reporting groups
Arm/Group | LUPRON | Placebo | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Full Range); unit: years] | 27.5 [20 to 35] | 28.25 [21 to 40] | 27.93 [20 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Anti-mullerian Hormone (AMH) Measured as a Continuous Variable, Specifically Assessing the Intra-person Change From Study Entry (Day 0) to 6-month Post-intervention Visit
Description: AMH was quantified in vitro a commercially available enzyme linked immunosorbent assay (ELISA) (Beckman Coulter; Marseille, France) was used for in vitro quantitative measurement of serum AMH.
Time Frame: Day 0 to 6-month post-intervention visit
Population: 8 subjects are listed in the breakdown of baseline characteristics. Samples were missing from one subject enrolled in the Placebo arm - therefore analysis throughout the majority of the reporting will include only 7 samples instead of 8 in the Placebo arm
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | LUPRON | Placebo
Number analyzed (Participants) | 6 | 7
ng/ml
  Baseline AMH (ng/ml) | 2.07 (1.92) | 3.87 (4.00)
  6 month AMH (ng/ml): number analyzed (Participants) | 5 | 1
  6 month AMH (ng/ml) | 0.72 (1.07) | 0.24 (0)

2. Secondary Outcome: Count of Patients With AMH of ≤1.0 ng/mL vs >1 ng/mL,
Description: AMH level ≤1.0 predicts onset of menopause within 5 years in normal women
Time Frame: baseline and 6 months
Population: 4 of the 7 subjects in the placebo arm dropped out of the study and 2 of the remaining subjects failed to have blood drawn at the 24 week (6 month) milestone, and 1 subject of the 6 subjects receiving active drug dropped out of the study before reaching the 24 week (6 month) milestone
Measure: Count of Participants; unit: Participants
Groups:
- PLACEBO: depot leuprolide acetate 3.75 mg: Monthly depot leuprolide acetate 3.75 mg vs placebo during cyclophosphamide administration. First dose of study drug given at least 10 days before following dose of cyclophosphamide if cyclophosphamide is given in biweekly or monthly boluses
Arm/Group | LUPRON | PLACEBO
Number analyzed (Participants) | 6 | 7
Participants
  Baseline AMH level ≤1.0 ng/ml | 3 | 6
  Baseline AMH level >1 ng/ml | 3 | 1
  6 Month AMH level ≤1.0 ng/ml: number analyzed (Participants) | 5 | 1
  6 Month AMH level ≤1.0 ng/ml | 4 | 1
  6 Month AMH level >1 ng/ml: number analyzed (Participants) | 5 | 1
  6 Month AMH level >1 ng/ml | 1 | 0

3. Secondary Outcome: Number of Participants With Either an AMH Level of >1 ng/mL OR Antral Follicle Count of >4.
Description: An AMH level of >1 ng/ml and/or an antral follicle count of >4 in either ovary is a strong predictor of residual ovarian function
Time Frame: baseline and 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LUPRON | PLACEBO
Number analyzed (Participants) | 6 | 7
Participants
  Baseline AMH >1 ng/ml or AFC>4 | 4 | 6
  6 Month AMH >1 ng/ml or AFC>4: number analyzed (Participants) | 5 | 1
  6 Month AMH >1 ng/ml or AFC>4 | 1 | 0

4. Secondary Outcome: Mean Antral Follicle Count (AFC)
Description: Mean antral follicle count (AFC) is the average number of follicles counted in each of 2 ovaries
Time Frame: baseline and 6 months
Population: 4 of the 7 subjects in the placebo arm dropped out of the study before reaching the 24 week (6 month) milestone, and 2 subjects of the 6 subjects receiving active drug did not have ultrasound performed at the 24 week (6 month) milestone
Measure: Mean (Standard Deviation); unit: # of ovarian follicles
Arm/Group | LUPRON | PLACEBO
Number analyzed (Participants) | 6 | 7
# of ovarian follicles
  Baseline Mean antral follicle count (AFC) | 10.3 (9.29) | 14.4 (12.4)
  6 Month Mean antral follicle count (AFC): number analyzed (Participants) | 4 | 3
  6 Month Mean antral follicle count (AFC) | 2.5 (1.29) | 17.7 (21.1)

5. Secondary Outcome: Mean Ovarian Volume.
Description: Mean ovarian volume reflects the preservation of ovarian tissue despite exposure to cyclophosphamide; reduced ovarian size is documented in cyclophosphamide treated patients
Time Frame: baseline and 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | LUPRON | PLACEBO
Number analyzed (Participants) | 6 | 7
cubic centimeters
  Baseline mean ovarian volume | 9.59 (2.69) | 7.68 (3.50)
  6 Month mean ovarian volume: number analyzed (Participants) | 4 | 3
  6 Month mean ovarian volume | 4.26 (1.93) | 6.97 (5.54)

ADVERSE EVENTS:
Time Frame: adverse events were collected from the time of randomization/baseline to the 6 month (24 week) follow up period The total interval of time for subjects in which AE's were collected spans approximately 6 months/24 weeks for each subject
Arm/Group | LUPRON | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/8
Other Adverse Events (participants affected / at risk) | 5/6 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUPRON (N=6) | Placebo (N=8)
clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Hospitalization for items listed below: (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — joint pain, shortness of breath, hypertension Classified as musculoskeletal because as the array of systems were all related to her systemic lupus and a lupus related flare of disease
Hospitalization for items listed below (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — joint pain, nausea, and hypertension, classified as musculoskeletal because as the array of systems were all related to her systemic lupus and a lupus related flare of disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUPRON (N=6) | Placebo (N=8)
leg striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hot flashes (Reproductive system and breast disorders) | 2 (2) | 4 (4)
hot and cold flashes (Reproductive system and breast disorders) | 0 (0) | 1 (1)
facial rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — this was not a lupus related rash
increased sweating (Reproductive system and breast disorders) | 0 (0) | 1 (1)
2 menstruations in 28 day cycle (Reproductive system and breast disorders) | 0 (0) | 1 (1)
fluid retention (Renal and urinary disorders) | 1 (1) | 0 (0)
worsening hypertension (Renal and urinary disorders) | 1 (1) | 0 (0) — this is felt to be secondary to the subject's fluid retention
bleeding at catheter site (Surgical and medical procedures) | 1 (1) | 0 (0) — hemodialysis catheter
pain in right hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain in right forearm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
stool incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
menstrual spotting in between cycles (Reproductive system and breast disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 0 (0) | 1 (1)
night sweats (Reproductive system and breast disorders) | 0 (0) | 1 (1)
bacterial overgrowth - GI related (Gastrointestinal disorders) | 0 (0) | 1 (1)
arthralgias (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
viral upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
edema of left calf, foot, and hand (Renal and urinary disorders) | 0 (0) | 1 (1)
pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes